CLINICAL TRIAL: NCT03068741
Title: Paramedic Initiated Treatment of Sepsis Targeting Out-of-hospital Patients (PITSTOP)
Acronym: PITSTOP
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Dr. Damon Scales (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Sunnybrook Research Institute (Other)
Responsible Party: Sponsor-Investigator, Dr. Damon Scales, MD, PhD, FRCPC, Sunnybrook Health Sciences Centre
Organization: Sunnybrook Health Sciences Centre (Other)
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: The PITSTOP RCT
Record Dates: First submitted 2017-02-06; First posted 2017-03-03 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Severe Sepsis or Septic Shock
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Ceftriaxone; Sodium Chloride; Injections

STUDY DESIGN:
Intervention Model Description: This is a 2x2 factorial RCT, with simultaneous randomization of individual patients into 2 randomized controlled trials.
  The first RCT compares administration of 1g of intramuscular ceftriaxone versus placebo. In this RCT, participants, care providers, investigators, and outcome assessors will all be masked to the treatment allocation.
  The second RCT compares a liberal fluid resuscitation (up to 2litres of intravenous 0.9% saline) versus conventional resuscitation (administration of intravenous 0.9% saline, started only when systolic blood pressure is <90mmHg and only continued until systolic blood pressure is >= 100mmHg). In this RCT, only participants and outcome assessors will be masked.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study drug and placebo are prepared in identical masked containers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Comparison 1: Prehospital Ceftriaxone (Active Comparator): 1g of Ceftriaxone will be administered by immediate intramuscular (IM) injection. The drug is provided in a sterile and completely covered vial as a white, odourless powder
  Interventions: Drug: Comparison 1: Prehospital Ceftriaxone
- Comparison 1: Placebo (Placebo Comparator): The placebo is provided in a sterile and completely covered vial.
  Interventions: Drug: Comparison 1: Placebo
- Comparison 2: Liberal fluids (Experimental): Paramedics will administer up to 2 litres of intravenous 0.9% saline solution to all participants in this arm regardless of blood pressure, reassessing for signs of volume overload after each 250ml.
  Interventions: Drug: Comparison 2: Liberal fluids
- Comparison 2: Conservative fluids (Active Comparator): Paramedics will administer 0.9% saline solution to participants who have systolic blood pressure <90mmHg, and will only continue the infusion until the systolic blood pressure is >=100mmHg.
  Interventions: Drug: Comparison 2: Conservative fluids

INTERVENTIONS:
Drug: Comparison 1: Prehospital Ceftriaxone — Paramedics will administer 1g of intramuscular ceftriaxone.
  Other Names: Ceftriaxone
  Arms: Comparison 1: Prehospital Ceftriaxone
Drug: Comparison 1: Placebo — Paramedics will administer an identical volume of reconstituted intramuscular placebo.
  Other Names: 0.9% saline for injection
  Arms: Comparison 1: Placebo
Drug: Comparison 2: Liberal fluids — Paramedics will administer up to 2 litres of intravenous saline (0.9%) to all patients regardless of systolic blood pressure, and reassessing this infusion after each 250ml are infused.
  Other Names: intravenous saline (0.9%) for injection
  Arms: Comparison 2: Liberal fluids
Drug: Comparison 2: Conservative fluids — Paramedics will administer intravenous saline (0.9%) according to the Medical Directive, which allows for infusion of fluids if systolic blood pressure is <90mmHg and continued until systolic blood pressure is >=100mmHg.
  Other Names: intravenous saline (0.9%) for injection
  Arms: Comparison 2: Conservative fluids

SUMMARY:
Sepsis occurs when a serious infection - most commonly infection of the lungs, urinary system, or blood - leads to acute organ failure. It is a common, expensive, and frequently lethal condition. A growing body of evidence suggests that early recognition and treatment of sepsis can improve survival.

Unfortunately, many patients with sepsis do not receive key therapies until physicians working in Emergency Departments have assessed them - often introducing marked delays. It is estimated that one-half of patients with sepsis are treated and transported to hospital by paramedics. This allows paramedics a unique opportunity to provide early treatment at the initial point of patient contact, thereby decreasing the time to treatment for these critically ill patients. This randomized controlled trial will evaluate whether prompt recognition followed by early antibiotics and/or intravenous fluids delivered by paramedics in the field leads to improved survival, compared to usual care, for patients who are transported to the hospital with sepsis.

DETAILED DESCRIPTION:
The ultimate goal of this research program is to evaluate a fundamental change in the delivery of sepsis care. Currently, patients with severe sepsis do not receive key evidence-based therapies until they have been assessed in emergency departments - often introducing considerable delays. This research tests whether integrating paramedics directly into a chain-of-survival for sepsis will improve outcomes for these critically ill patients. In essence, this research seeks to break down silos of care, delivering sepsis treatments based on when they are needed, rather than on where the patient is physically located. If the trial is positive, the results will have broad implications for other health systems by showing that prehospital identification and treatment of sepsis increases the number of patients that survive this life-threatening condition. If the trial fails to demonstrate effectiveness of prehospital sepsis treatments, it will ensure that resources are not needlessly invested in large-scale implementations of paramedic sepsis protocols, as has been done in several other jurisdictions. A lack of benefit would also cast doubt on the observational data suggesting that early antibiotics are important, and suggest a more restrained approach to empiric antibiotic therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Sepsis, defined as (all 3 must be present): i) Paramedic suspects possible infection: e.g. suspected pneumonia, urinary tract infection, skin infection, bone and joint infection, intra-abdominal infection, meningitis ii) Presence of fever: Temperature ≥ 38.0°C measured by paramedic or history of fever during previous 24 hours iii) Presence of hypotension: Systolic blood pressure < 100mmHg
2. Age ≥ 18 years

Exclusion Criteria:

1. Post cardiac arrest
2. Suspected ST-segment elevation myocardial infarction (STEMI)
3. Suspected acute cerebrovascular accident (CVA)
4. Acute severe trauma
5. Obvious severe non-traumatic bleeding
6. Signs of fluid overload
7. Suspected acute congestive heart failure (CHF)
8. Known Clostridium difficile infection within the last 6 weeks
9. Known pregnancy or breastfeeding
10. Known allergy or sensitivity to penicillin or cephalosporin
11. Known to be receiving oral or subcutaneous anticoagulants or low molecular weight heparin
12. Paramedic is unable to identify patient by first and last name and/or health card number

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2040 (Estimated)
Dates: Start 2020-03-23 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Primary outcome: mortality prior to hospital discharge to day 90. | 90 days
  Dichotomous outcome reported as percentage

SECONDARY OUTCOMES:
Mortality at 90 days after enrollment | 90 days after enrollment
  Dichotomous outcome reported as percentage
Organ dysfunction during first 24 hours (mechanical ventilation, vasopressor therapy (any), dialysis | 24 hours
  Dichotomous outcome reported as percentage
Organ dysfunction during hospitalization (mechanical ventilation) | until hospital discharge, measured up to maximum of day 90
  Dichotomous outcome reported as percentage
duration of hospital admission (if any) | until hospital discharge, measured up to maximum of day 90
  Measured in days from time of randomization
duration of first ICU admission (if any) | until ICU discharge, measured up to maximum of day 90
  Measured in days from time of randomization
Proportion of patients with positive blood cultures obtained in hospital | 24 hours
  Dichotomous outcome reported as percentage
Microbiology results (if any) | 24 hours
  Descriptive outcome, reported as frequency distribution of positive culture results
Proportion of patients receiving antibiotics within first 24 hours of hospitalization | 24 hours
  Dichotomous outcome reported as percentage
Frequency distribution and mean time to first dose of antibiotics (if any) within first 24 hours of hospitalization | 24 hours
  Measured in hours from time of randomization
Proportion of patients receiving IV fluids (>250mL) within first 24 hours of hospitalization | 24 hours
  measured in milliliters
Total amount of IV fluids administered during transport and first 24 hours of hospitalization (if any) | 24 hours
  measured in milliliters
Proportion of patients with pulmonary edema identified during transport to hospital and on initial chest x-ray | during transport and on initial chest x-ray (if completed)
  Dichotomous outcome reported as percentage
Proportion of patients with blood, urine, sputum cultures that grow organisms resistant to ceftriaxone | 24 hours
  Dichotomous outcome reported as percentage
Proportion of patients diagnosed with sepsis or infection by emergency department physician | during admission
  Dichotomous outcome reported as percentage
Proportion of hospitalized patients who grow any antibiotic-resistant organism (methicilin resistant S. aureus, Clostridium difficile, extended beta-lactamase resistant organisms) | during admission
  Dichotomous outcome reported as percentage
Proportion of patients with anaphylaxis or suspected allergic reactions to study medication | during admission
  Dichotomous outcome reported as percentage

CONTACTS AND LOCATIONS:
Overall Officials: Damon Scales, MD PhD FRCPC, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (4):
- Canada (4):
  - Halton Region Paramedic Services, Toronto, Ontario
  - Peel Region Paramedic Services, Toronto, Ontario
  - Toronto Paramedic Services, Toronto, Ontario
  - York Region Paramedic Services, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Scales DC, Rogowsky A, Burry L, Christenson J, Daneman N, Drennan IR, Hillier M, Jenneson S, Klein G, Mazzulli T, Moran P, Morris AM, Morrison LJ, Pinto R, Rubenfeld GD, Seymour CW, Stenstrom R, Verbeek PR, Cheskes S. Prehospital antibiotics and intravenous fluids for patients with sepsis: protocol for a 2x2 factorial randomised controlled trial. BMJ Open. 2025 May 27;15(5):e104257. doi: 10.1136/bmjopen-2025-104257. PMID 40436458